CLINICAL TRIAL: NCT01377805
Title: Head Circumference Growth in Children Who Develop Multiple Sclerosis Later in Life -- a Retrospective Analysis
Brief Title: Head Circumference Growth in Children Who Develop Multiple Sclerosis Later in Life
Status: Withdrawn | Type: Observational
Why Stopped: No participants
Sponsor: Genetic Disease Investigators (Other)
Responsible Party: Sponsor
Other Study IDs: 61/3529
Record Dates: First submitted 2011-06-19; First posted 2011-06-21 (Estimated); Last update posted 2024-02-14 (Actual); Status verified 2015-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis hydrocephalus
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Multiple Sclerosis patients: Multiple sclerosis patients

SUMMARY:
Multiple sclerosis patients commonly develop generalized ventricular dilation with or without cerebral atrophy over time. Case studies in the literature have noted some multiple sclerosis patients develop the typical "normal pressure hydrocephalus" triad of dementia, gait disturbance and incontinence which were responsive to shunts.

Many patients with connective tissue disorders (Ehlers-Danlos Syndrome) develop Multiple Sclerosis and studies indicate that in the Multiple Sclerosis population, there exists over 10% more Ehlers-Danlos patients than in the normal population.

Because studies are indicating a form of external communicating hydrocephalus in the Ehlers-Danlos population, the author hypothesizes the same type of hydrocephalus may occur in the Multiple Sclerosis population.

To evaluate this hypothesis, investigators will retroactively evaluate the head circumference of Multiple Sclerosis patients between birth and 15 months (before the skull sutures have closed).

DETAILED DESCRIPTION:
Multiple sclerosis patients commonly develop generalized ventricular dilation with or without cerebral atrophy over time. Case studies in the literature have noted some multiple sclerosis patients develop the typical "normal pressure hydrocephalus" triad of dementia, gait disturbance and incontinence which were responsive to shunts.

Many patients with connective tissue disorders (Ehlers-Danlos Syndrome) develop Multiple Sclerosis and studies indicate that in the Multiple Sclerosis population, there exists over 10% more Ehlers-Danlos patients than in the normal population.

Because studies are indicating a form of external communicating hydrocephalus in the Ehlers-Danlos population, the author hypothesizes the same type of hydrocephalus may occur in the Multiple Sclerosis population.

To evaluate this hypothesis, investigators will retroactively evaluate the head circumference of Multiple Sclerosis patients between birth and 15 months (before the skull sutures have closed).

High pressure on the brain (even if subtle) could be evidence of congenital CCSVI (cerebrospinal venous insufficiency), increased cerebrospinal fluid (CSF) production, the poor drainage of cerebral spinal fluid, or a combination of all. Retrospective examination of skull expansion is a necessary step to ascertain these possibilities, allowing for early treatment and the hope of avoidance of the neurological symptoms, and often disabling effects. It is the author's belief that "Benign External Hydrocephalus" is not a benign condition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Sclerosis

Exclusion Criteria:

* Excludes CIS (clinically isolated syndrome)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Multiple Sclerosis, no geographic limitations
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Measurement of Head Circumference in Multiple Sclerosis patients (retrospectively) | Retrospectively, between patient's birth to 15 months of age
  Measurement of head circumferences, weight and length of children (retrospectively), will be compared to "normals" as established by the U.S. Department of Health and Human Services, Centers for Disease Control and Prevention (CDC), 2008.

CONTACTS AND LOCATIONS:
Overall Officials: Diana L Driscoll, O.D., Principal Investigator — Genetic Disease Investigators
Locations (1):
- POTS Care, Colleyville, Texas, United States

REFERENCES:
- [Background] O'Brien T, Paine M, Matotek K, Byrne E. Apparent hydrocephalus and chronic multiple sclerosis: a report of two cases. Clin Exp Neurol. 1993;30:137-43. PMID 7712624
- [Background] Vilisaar J, Harikrishnan S, Suri M, Constantinescu CS. Ehlers-Danlos syndrome and multiple sclerosis: a possible association. Mult Scler. 2008 May;14(4):567-70. doi: 10.1177/1352458507083187. Epub 2008 Jan 21. PMID 18208891